CLINICAL TRIAL: NCT02647762
Title: A Phase 3, Randomized, Double-Blind, Active- and Placebo-controlled, Parallel-group Trial to Evaluate the Efficacy and Safety of CF101 Compared to Methotrexate in the Treatment of Early Rheumatoid Arthritis
Brief Title: CF101 Therapy Compared to Methotrexate Therapy for Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis results
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-301RA
Record Dates: First submitted 2015-12-16; First posted 2016-01-06 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CF101 1mg (Experimental): CF101 1mg, orally q12 hours
  Interventions: Drug: CF101 1 mg
- CF101 2mg (Experimental): CF101 2mg, orally q12 hours
  Interventions: Drug: CF101 2 mg
- MTX once weekly (Active Comparator): MTX 5 mg tablets, given once weekly at 10 mg/week (2 tablets) for the first 2 weeks, then 15 mg/week (3 tablets) for the next 2 weeks, then 20 mg/week (4 tablets) thereafter.
  Interventions: Drug: MTX
- Placebo (Placebo Comparator): Placebo control , orally q12 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF101 1 mg — CF101 tablets, 1mg BID for 12 weeks
  Other Names: IB-MECA; Piclidenosone
  Arms: CF101 1mg
Drug: CF101 2 mg — CF101 tablets, 2 mg BID for 12 weeks
  Other Names: IB-MECA; Piclidenosone
  Arms: CF101 2mg
Drug: Placebo — Placebo tablets, 1mg BID for 12 weeks
  Arms: Placebo
Drug: MTX — MTX 5 mg tablets, given once weekly at 10 mg/week (2 tablets) for the first 2 weeks, then 15 mg/week (3 tablets) for the next 2 weeks, then 20 mg/week (4 tablets) thereafter, for 12 weeks.
  Arms: MTX once weekly

SUMMARY:
This trial will test the hypothesis that the administration of CF101, a novel anti-inflammatory agent, to patients with rheumatoid arthritis will relieve signs and symptoms of the disease. CF101 effect will be in comparison to MTX in this study population.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, active- and placebo-controlled, parallel-group study in subjects with clinically active RA but who are MTX-naïve. Subjects who meet enrollment criteria will be randomized to 1 of 4 groups in a 2:2:2:1 ratio: CF101 1 mg, CF101 2 mg, MTX, or matching placebo tablets. CF101 or matching placebo will be administered every 12 hours for up to 24 weeks on treatment. MTX or matching placebo will be administered once a week Screening examinations will occur within 6 weeks prior to dosing. The following conventional drugs for RA treatment must be stable for the respective designated periods prior to the Screening Visit and must remain so during protocol participation: nonsteroidal anti-inflammatory drugs (NSAIDS), and corticosteroids for >1 month. All subjects will receive oral folate (minimum dose 5 mg/week) or oral folinic acid (up to 10 mg/week), based on the Investigator's preference.

Disease activity will be assessed using swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and CRP. Efficacy will be assessed by Disease Activity Score 28 using the erythrocyte sedimentation rate (DAS28-ESR), ACR response criteria and European League Against Rheumatism (EULAR) response criteria : swollen and tender joint counts, physician global assessment (by visual analog scale, patient global assessment , patient reported pain, a Health Assessment Questionnaire (HAQ) Disability Index (DI) , Westergren ESR levels, and CRP levels. Assessments will occur at Screening, Baseline (Week 0), and Weeks 4, 8, 12 16, 20, and 24. At Weeks 12, 16, and 20, any subject who has not experienced at least 20% improvement in both the number of swollen and number of tender joints will be given rescue therapy with open-label oral MTX and followed through Week 24.

PK will be assessed in a subgroup of approximately 100 subjects at Week 0, Week 8, and Week 12. All subjects in the PK cohort will have samples collected for PK at time 0, and each subject will have additional samples drawn at 2 of the following post-dose time points: 1, 2, 3, 4, 6, and 8 hours. Whole blood sample for A3AR expression will be assessed in approximately 100 subjects at selected sites at Screening and Week 12, or end of dosing, if occurring before Week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 18-75 years.
2. Meet the criteria of the American College of Rheumatology for RA (Arnett FC et al. Arthritis Rheum 1988;31:315-324, Appendix 1).
3. Not bed- or wheelchair-bound.
4. Active RA, as indicated by EULAR Disease Activity Score (Fransen, vanRiel, 2005, DAS28, 2015) (DAS28) >3.2.
5. Demonstrate at least 6 swollen and at least 6 tender joints.
6. If taking an NSAID, dose has been stable for at least 1 month prior to the Screening Visit, and will remain unchanged during protocol participation.
7. If taking an oral corticosteroid, dose is <10 mg/day prednisone or equivalent, has been stable for at least 1 month prior to the Screening Visit, and will remain unchanged during protocol participation.
8. In the Investigator's opinion, the ability to understand the nature of the study and any hazards of participation, and to communicate satisfactorily with the Investigator and to participate in, and to comply with, the requirements of the entire protocol.
9. Negative Screening serum pregnancy test for female subjects of childbearing potential.
10. Females of childbearing potential must utilize, throughout the course of the trial, 2 methods of contraception deemed adequate by the Investigator (for example, oral contraceptive pills plus a barrier method).
11. All aspects of the protocol explained and written informed consent obtained.

Exclusion Criteria:

1. Prior receipt of MTX.
2. Prior receipt of >1 regimen of synthetic small-molecule DMARDs.
3. Receipt of any non-MTX synthetic small-molecule DMARDs (including but not limited to sulfasalazine, chloroquine/hydroxychloroquine, azathioprine, and/or leflunomide) for at least 1 month prior to the Screening Visit or concomitantly during the trial.
4. Receipt of tofacitinib at any time during the 4-week period prior to the Screening Visit or concomitantly during the trial.
5. Receipt of a biologic anti-rheumatic agent (including, but not limited to, etanercept, abatacept, infliximab, golimumab, adalimumab, tocilizumab, certolizumab, and rituximab) at any time prior to or concomitantly during the trial.
6. Levels of rheumatoid factor (RF) and anti-cyclic citrullinated peptide (CCP) antibody that are both >3 times the upper limit of the laboratory normal value at the Screening Visit.
7. Receipt of parenteral or intra-articular corticosteroids during the 1 month prior to the Screening Visit.
8. Participation in a previous trial CF101 trial.
9. Presence or history of uncontrolled arterial hypertension or symptomatic hypotension.
10. Heart disease which is, in the Investigator's judgment, clinically significant or unstable, including coronary artery disease, congestive heart failure, uncontrolled arrhythmia, or other significant findings on Screening electrocardiogram (ECG).
11. Clinical laboratory abnormalities at the Screening Visit as follows:

    1. Hemoglobin level <9.0 gm/dL
    2. Platelet count <125,000/mm3
    3. White blood cell (WBC) count <3000/mm3
    4. Serum creatinine level outside the central laboratory's normal limits
    5. Liver aminotransferase (ALT and/or AST) levels greater than 2 times the central laboratory's upper limit of normal.
12. Known or suspected immunodeficiency or human immunodeficiency virus positivity.
13. Pregnancy, lactation, or inadequate contraception as judged by the Investigator.
14. Participation in another investigational drug or vaccine trial concurrently or within 30 days prior to Screening.
15. Active drug or alcohol dependence.
16. History of malignancy within the past 2 years (excluding excised basal or squamous cell carcinoma of the skin).
17. Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of oral CF101, BID for 12 weeks to subjects with active rheumatoid arthritis (RA) relative to oral methotrexate (MTX) as assessed by the proportion of subjects achieving a Disease Activity Score (DAS) of Low Disease Activity (LDA) | 12 weeks
  Proportion of subjects achieving Disease Activity Score (DAS) (based on Erythrocyte Sedimentation Rate) of Low Disease Activity (<3.2, where lower scores indicate lower disease activity) at Week 12
Assess the adverse event profile of daily oral CF101 under the conditions of the trial | 24 weeks
  Nature, incidence and severity of treatment-emergent adverse events (TEAEs)
Describe the pharmacokinetics (PK) of CF101 under the conditions of the trial | 24 weeks
  Plasma CF101 levels will be determined

SECONDARY OUTCOMES:
Determine the efficacy of oral CF101 when administered daily for 24 weeks to subjects with active RA relative to oral MTX, as assessed by the proportion of subjects achieving DAS remission | 24 weeks
  Change and percent change from baseline in DAS28
Explore the relationship between whole blood adenosine A3 receptor (A3AR) expression and treatment response | 24 weeks
  A3AR expression will be assessed on whole blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma
Locations (35):
- Bosnia and Herzegovina (5):
  - Can-Fite Investigational Site #252, Banja Luka
  - Can-Fite Investigational Site #256, Banja Luka
  - Can-Fite Investigational Site #253, Mostar
  - Can-Fite Investigational Site #251, Sarajevo
  - Can-Fite Investigational Site #255, Tuzla
- Can-Fite Investigational Site #751, Barrie, Canada
- Israel (2):
  - Can-Fite Investigational Site #309, Ashkelon
  - Can-Fite Investigational Site #302, Haifa
- Moldova (3):
  - Can-Fite Investigational Site #581, Chisinau
  - Can-Fite Investigational Site #582, Chisinau
  - Can-Fite Investigational Site #583, Chisinau
- Poland (3):
  - Can-Fite Investigational Site #401, Bialystok
  - Can-Fite Investigational Site #402, Bochnia
  - Can-Fite Investigational Site #403, Poznan
- Romania (12):
  - Can-Fite Investigational Site #559, Brăila
  - Can-Fite Investigational Site #551, Bucharest
  - Can-Fite Investigational Site #552, Bucharest
  - Can-Fite Investigational Site #553, Bucharest
  - Can-Fite Investigational Site #562, Bucharest
  - Can-Fite Investigational Site #564, Bucharest
  - Can-Fite Investigational Site #565, Bucharest
  - Can-Fite Investigational Site #558, Constanța
  - Can-Fite Investigational Site #563, Craiova
  - Can-Fite Investigational Site #561, Iași
  - Can-Fite Investigational Site #555, Oradea
  - Can-Fite Investigational Site #554, Timișoara
- Serbia (9):
  - Can-Fite Investigational Site #212, Belgrade
  - Can-Fite Investigational Site #223, Bor
  - Can-Fite Investigational Site #219, Kragujevac
  - Can-Fite Investigational Site #215, Niš
  - Can-Fite Investigational Site #213, Novi Sad
  - Can-Fite Investigational Site #222, Pirot
  - Can-FIte Investigational Site #221, Sremska Mitrovica
  - Can-Fite Investigational Site #214, Šabac
  - Can-Fite Investigational Site #220, Zrenjanin